CLINICAL TRIAL: NCT03558178
Title: The Effectiveness and Cost-effectiveness of Doin (Conduction Exercise) for Chronic Neck Pain: A Multi-center Randomized Controlled Trial
Brief Title: The Effectiveness and Cost-effectiveness of Doin (Conduction Exercise) for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2018-03
Record Dates: First submitted 2018-06-01; First posted 2018-06-15 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doin with Acupuncture (Experimental): An acupuncture physician will administer acupuncture at a total 6-12 acupoints in the upper and middle trapezius areas (mandatory points: both SI15, TE15, and LI16; and selective points: GB20, BL10, GV14, SI14, and Hyeopcheok (Huatuo Jiaji, EX B2) points at C3-5 levels). Cervical Doin (conduction exercise) will be performed with the needles in situ by increasing the cervical range of motion (rotation) with physician guidance and isometric resistance exercise as indicated.
  Interventions: Procedure: Doin with acupuncture; Device: Acupuncture
- Acupuncture (Active Comparator): An acupuncture physician will administer acupuncture at a total 6-12 acupoints in the upper and middle trapezius areas (mandatory points: both SI15, TE15, and LI16; and selective points: GB20, BL10, GV14, SI14, and Hyeopcheok (Huatuo Jiaji, EX B2) points at C3-5 levels).
  Interventions: Device: Acupuncture

INTERVENTIONS:
Procedure: Doin with acupuncture — Doin (conduction exercise) will be performed with the needles in situ by increasing the cervical range of motion (rotation) with physician guidance and isometric resistance exercise as indicated. Doin sessions will be conducted 2 times a week for 5 weeks (total 10 sessions).
  Other Names: Doin Exercise with acupuncture; Do-in Exercise with acupuncture; Conduction Exercise with acupuncture
  Arms: Doin with Acupuncture
Device: Acupuncture — Acupuncture will be performed with manual stimulation (needle twirling) to evoke de-qi sensation. Acupuncture sessions will be conducted 2 times a week for 5 weeks (total 10 sessions).

SUMMARY:
A multi-center randomized controlled trial assessing the comparative effectiveness and cost-effectiveness of Doin (conduction exercise) with acupuncture for chronic neck pain

DETAILED DESCRIPTION:
A multi-center randomized controlled, parallel, assessor-blinded full-scale trial will be conducted based on the results of the pilot study to evaluate the comparative clinical effectiveness and cost-effectiveness of Doin (conduction exercise) with acupuncture for chronic neck pain patients compared to acupuncture alone as assessed using pain, functional disability, health-related quality of life, economic evaluation, and safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Neck area pain duration of 6 months or longer
* Current Numeric Rating Scale (NRS) for neck area pain of 5 or higher
* Patients who have agreed to voluntarily participate in the clinical trial and given written informed consent

Exclusion Criteria:

* Patients diagnosed with serious pathology(s) which may cause neck pain (e.g. malignant tumor, spinal infection, inflammatory spondylitis)
* Progressive neurologic deficit or severe neurologic symptoms (e.g. cauda equina syndrome, progressive muscle weakness)
* Pathologies of non-spinal or soft tissue origin or high severity which may cause neck or radiating arm pain (e.g. malignant tumor, spinal infection, inflammatory spondylitis, fibromyalgia, rheumatic arthritis, gout)
* Other chronic diseases which may interfere with treatment effect or interpretation of results (e.g. cardiovascular disorder, renal disease, diabetic neuropathy, dementia, epilepsy)
* Current intake of steroids, immunosuppressant medicine, psychiatric medicine or other medication which may interfere with treatment results
* Patients considered unsuitable or unsafe to receive acupuncture (e.g. patients with hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine intake, severe diabetes with high risk of infection, severe cardiovascular diseases)
* Patients who were treated with invasive interventions such as acupuncture or injections, or with medicine that may potentially influence pain such as NSAIDs (nonsteroidal antiinflammatory drugs) within the past week
* History of cervical surgery within the past 3 months
* Pregnancy or plans of pregnancy
* Severe psychopathy
* Participation in other clinical studies
* Inability to give written informed consent
* Other reasons rendering trial participation inappropriate as judged by the researchers

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Difference between visual analogue scale (VAS) of neck pain for the past 3 days at 5 weeks post-baseline and baseline | Week 5 post-baseline (screening)
  VAS uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain' and 'worst pain possible' (labels may vary by study). Scores are recorded in millimeters with a total range of 0-100 millimeters.

SECONDARY OUTCOMES:
Difference between visual analogue scale (VAS) of radiating arm pain for the past 3 days at each timepoint and baseline, respectively | Week 1, 2, 3, 4, 5, 6 post-baseline (screening)
  VAS uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain' and 'worst pain possible' (labels may vary by study). Scores are recorded in millimeters with a total range of 0-100 millimeters.
Difference between numeric rating scale (NRS) of neck pain for the past 3 days at each timepoint and baseline, respectively | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Difference between numeric rating scale (NRS) of radiating arm pain for the past 3 days at each timepoint and baseline, respectively | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Difference between Neck Disability Index (NDI) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The NDI evaluates functional impairment and is a 10-item questionnaire developed to assess the level of disability due to neck pain. Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to neck pain.
Difference between Northwick Park Neck Pain Questionnaire (NPQ) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The NPQ evaluates functional impairment for the past 3 days in this study and is a patient reported outcome of subjective neck pain and pain reduction. The NPQ is a 9-item questionnaire developed to assess the level of disability due to neck pain. Each item is graded into 5 levels, each representing a score of 0-4. Higher scores indicate greater limitation relating to neck pain.
Patient Global Impression of Change (PGIC) | Week 6, Month 3, 6, 9, 12 post-baseline (screening)
  PGIC grades the level of subjective improvement into 7 levels (1, very much improved; 2, much improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; and 7, very much worse).
Physical examination | Week 1, 6 post-baseline (screening)
  Pain upon movement in cervical range of motion (ROM) will be assessed.
Difference between the 5 level version of EuroQol-5 Dimension (EQ-5D-5L) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  EQ-5D is a tool developed for health-related quality of life (HRQoL) assessment, and is widely used in the health care sector. Scores range from -1, 'health worse than death' to 1, 'perfect health'. EQ-5D-5L has 5 dimensions covering current health status and functionality: mobility (M), self care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD), to be rated out of 5 grades (1, no problem; 2, slight problem; 3, some/moderate problem; 4, severe problem; 5, extreme problem).
Difference between the EuroQol Visual Analogue Scale (EQ-VAS) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  EQ-VAS uses a vertical 10cm line labeled at each end with scale anchors. EQ-VAS is used to indicate the patient's health state and patients are asked to mark a point that represents their health state between the anchors of 'worst health state' and 'best health state imaginable'. Scores are recorded in millimeters with a total range of 0-100 millimeters.
Difference between the Short Form Health Survey 12 (SF-12) at each timepoint and baseline, respectively | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  SF-12 is a simplified version of SF-36. SF-12 assesses health-related quality of life (HRQoL) across 8 domains with 1-2 items per domain: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Higher scores indicate better HRQoL.
Economic evaluation (medical costs) | Week 1, 6, Month 3, 6, 9, 12 post-baseline (screening)
  Economic evaluation of medical costs will be performed to assess cost-effectiveness of the 2 groups.
Economic evaluation (time-related costs) | Week 2 post-baseline (screening)
  Economic evaluation of time-related costs will be performed to assess cost-effectiveness of the 2 groups.
Economic evaluation (lost productivity costs) | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  Economic evaluation of lost productivity costs will be performed to assess cost-effectiveness of the 2 groups.
Credibility and Expectancy Questionnaire | Week 1 post-baseline (screening)
  The credibility and expectancy questionnaire will be used to assess treatment expectation on a 9-point Likert scale. Participants will be asked to select an answer to the following questions on their first visit of Week 1 (1='not at all'; and 5='somewhat'; to 9='very much'): "How much do you expect that treatment will alleviate your symptoms during the study period?"
Drug Consumption (drug type) | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The drug type of prescription intake for medicine or rescue medicine (acetaminophen) will be recorded.
Drug Consumption (drug dose) | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The drug dose of prescription intake for medicine or rescue medicine (acetaminophen) will be recorded.
Other treatments (treatment type) | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The type of other treatments received (e.g. physical therapy, injections) will be recorded.
Other treatments (treatment frequency) | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening)
  The frequency of other treatments received (e.g. physical therapy, injections) will be recorded.
Adverse events | Week 1, 2, 3, 4, 5, 6, Month 3, 6, 9, 12 post-baseline (screening) (every visit)
  Physicians will monitor and record any unexpected or unintended patient reaction to Chuna or usual care at each visit. Adverse events (AEs) associated with Chuna will include, but not be limited to, AEs anticipated from previous reports of manual therapy, and will stay open to all possibilities taking into consideration other potential, unknown AEs.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, Ph.D, Principal Investigator — Jaseng Medical Foundation
Locations (5):
- South Korea (5):
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi-do
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul
  - Kyung Hee University Oriental Medicine Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SM, Kim SJ, Nam D, Park YC, Kim EJ, Ha IH, Lee YJ. Comparison of preference-based health-related quality of life measures for chronic neck pain: a pooled analysis of data from three RCTs. BMJ Open. 2024 Dec 26;14(12):e086104. doi: 10.1136/bmjopen-2024-086104. PMID 39725423
- [Derived] Lee SH, Lee J, Lee YJ, Kim MR, Cho JH, Kim KW, Ha IH. Effectiveness and cost-effectiveness of acupuncture with Doin therapy for chronic neck pain: a study protocol for a multicentre, randomised controlled clinical trial. BMJ Open. 2019 May 10;9(5):e026632. doi: 10.1136/bmjopen-2018-026632. PMID 31079083